CLINICAL TRIAL: NCT04627025
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Apraglutide in Adult Subjects With Short Bowel Syndrome and Intestinal Failure (SBS-IF)
Brief Title: Trial to Evaluate Efficacy and Safety of Apraglutide in SBS-IF
Acronym: STARS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VectivBio AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA799-007; 2020-001202-32 (EudraCT Number)
Record Dates: First submitted 2020-10-22; First posted 2020-11-13 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel Syndrome; Intestinal Failure; SBS; SBS-IF; GLP-2; Short Bowel Syndrome Intestinal Failure
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure | interventions — apraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apraglutide SC injections, once weekly (Experimental): Peptide analogue of GLP-2
  Interventions: Drug: apraglutide
- Placebo (Placebo Comparator): Placebo for apraglutide, SC injection once weekly
  Interventions: Drug: apraglutide

INTERVENTIONS:
Drug: apraglutide — Apraglutide is a peptide analogue of GLP-2 under development for treatment of SBS-IF, which acts as a full agonist at the GLP-2 receptor with in vitro potency and selectivity comparable with native GLP-2.

SUMMARY:
The primary objective of the trial is the confirmation of the efficacy of apraglutide to evaluate the efficacy of weekly subcutaneous apraglutide in reducing parenteral support dependency.

DETAILED DESCRIPTION:
This is an international, multicenter, double-blind, randomized, placebo-controlled, trial to evaluate the efficacy and safety of weekly SC injections of apraglutide in adult subjects with SBS-IF. The active pharmaceutical ingredient is apraglutide, a GLP-2 analogue.

The trial consists of a screening phase, a treatment phase of 48 weeks, and a safety follow-up phase. Trial participants will receive, after successful screening, once weekly apraglutide.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent for this trial prior to any trial specific assessment.
2. Male and female subjects with SBS-IF, receiving parenteral support (PS), secondary to surgical resection of the small intestine with either stoma or colon-in-continuity (CIC).
3. Subject must require PS at least 3 days per work and be considered stable.
4. No restorative surgery intended to change PS requirements in the trial period.
5. Age ≥18 years at screening.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Major abdominal surgery in the last 6 months prior to screening.
3. History of cancer (including colon carcinoma) or clinically significant lymphoproliferative disease within ≤5 years, except for adequately treated basal cell skin cancer.
4. Evidence of active inflammatory GI conditions in the previous 6 months.
5. Evidence of decompensated heart failure.
6. Evidence of severe renal or hepatic impairment.
7. Any previous use of growth factors such as growth hormone (GH), native GLP-2, GLP-1, or GLP-2 or GLP-1 analogues should be discussed with the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in actual weekly PS volume at Week 24. | At week 24 of treatment

SECONDARY OUTCOMES:
Subjects who achieve a reduction of at least 1 day per week of PS at Weeks 24 / 48 (CIC only). | Weeks 24 and 48 of treatment
Relative change from baseline in actual weekly PS volume at Weeks 12 / 24 / 48 (CIC only). | Weeks 12 / 24 / 48 of treatment
Subjects reaching enteral autonomy at Weeks 24 / 48 (CIC only). | Weeks 24 / 48 of treatment
At least 20% reduction of PS volume from baseline at Weeks 20 / 24. | Weeks 20 / 24 of treatment
Calorie reduction in the PN at Weeks 24. | Weeks 24 of treatment
Change from baseline on the Pittsburgh Sleep Quality Inventory (PSQI) at Weeks 24 / 48 (CIC only) | Weeks 24 / 48 of treatment
Change from baseline on the Patient Global Impression of Change (PGIC) at Weeks 24 / 48 (CIC only) | Weeks 24 / 48 of treatment.
Change from baseline on the Patient Global Impression of Treatment Satisfaction (PGI-TS) at week 24 and 48 (CIC only). | Weeks 24 / 48 of treatment
Change from baseline on the Patient Global Impression of Satisfaction with Parenteral Support (PGI-SPS) at Week 24 and 48 (CIC only). | Weeks 24 / 48 of treatment
Change from baseline on the Patient Global Impression of Parenteral Support Impact (PGI-PSI) at Week 24 and 48 (CIC only). | Weeks 24 / 48 of treatment
Absorption rate constant (ka) of apraglutide through population PK data analysis | Weeks 0 / 24 of treatment
Apparent clearance (CL/F) of apraglutide through population PK data analysis | Weeks 0 / 24 of treatment
Apparent volume of distribution (Vz/F) of apraglutide through population PK data analysis | Weeks 0 / 24 of treatment
At least 40% reduction of PS volume at Weeks 20 and 24 (Stoma only) | Weeks 20 / 24 of treatment
Trough plasma concentrations (Ctrough) at every other visit during the prolonged dosing period (CIC only) | Weeks 24 / 48 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (68):
- United States (13):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Gastroenterology Group of Naples, Naples, Florida
  - Northwestern University, Chicago, Illinois
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Center for Human Nutrition, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington
- University Hospital Foundation Favaloro, Buenos Aires, Argentina
- Belgium (2):
  - Universitair Ziekenhuis Leuven - Gasthuisberg, Leuven, Vlaams Brabant
  - University Hospital Brussels, Brussels
- Czechia (6):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Hospital Novy Jicin, Nový Jičín
  - University Hospital Plzen, Pilsen
  - University Hospital Kralovske Vinohrady, 2nd Internal Clinic, Prague
  - General University Hospital in Prague, Prague
- Rigshospitalet - University Hospital Copenhagen, Copenhagen, Denmark
- France (6):
  - Hôpital Beaujon, Clichy
  - CHU Hôtel Dieu, Nantes
  - Hôpital ARCHET II, Nice
  - Hôpital Haut-Lévèque, Pessac
  - Hospices Civils de Lyon, Pierre-Bénite
  - Brabois Adults Hospital, Vandœuvre-lès-Nancy
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Hospital Bonn, Bonn
  - Asklepios Klinik St. Georg, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Muenster, Münster
- Hungary (4):
  - Medical Centre, Hungarian Defence Forces, Budapest
  - Semmelweis University, Budapest
  - St. Imre University Teaching Hospital Budapest, Budapest
  - University of Szeged, Szeged
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Polyclinic S. Orsola-Malpighi, Bologna
  - University Polyclinic Foundation "Agostino Gemelli" - IRCCS, Rome
  - Citta della salute e della Scienza di Torino Hospital, Torino
- Japan (5):
  - Yokohama Municipal Citizen's Hospital, Kanagawa
  - Yokohama City University Medical Center, Kanagawa
  - National University Corportation Tohoku University Tohoku University Hospital, Miyagi
  - Osaka University Hospital, Osaka
  - JCHO Tokyo Yamate Medical Center, Tokyo
- Alesund Hospital, Ålesund, Norway
- Poland (5):
  - Stadmedica, Non-Public Healthcare Facility, Bydgoszcz
  - COPERNICUS Limited Liability Company, Gdansk
  - M. Pirogow Provincial Specialized Hospital, Lodz
  - Gastromed Poland Sp. z o.o., Lublin
  - Stanley Dudrick Multispecialty Hospital, Skawina
- South Korea (3):
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Soeul
  - Samsung Medical Center, Soeul
- Spain (3):
  - University General Hospital Gregorio Maranon, Madrid
  - University Hospital 12 de Octubre, Madrid
  - University Hospital Virgen del Rocio, Seville
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Far Eastern Memorial Hospital, New Taipei City, Taiwan
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - St Mark's Hospital, Harrow
  - Royal London Hospital, London
  - University College Hospital, London
  - Salford Royal Hospital, Salford